CLINICAL TRIAL: NCT03629522
Title: Effects on Ondansetron on Maternal Hemodynamics After Cesarean Section Under Spinal Anesthesia: a Randomized Controlled Trial
Brief Title: Effects of Ondansetron on Hemodynamics in Cesarean Section Under Spinal Anesthesia
Acronym: EffOnd
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Mahdia (Other)
Responsible Party: Principal Investigator, Majdoub Ali MD, clinical professor, University Hospital, Mahdia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C/SOP2018
Record Dates: First submitted 2018-04-24; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Ondansetron; Cesarean Section; Spinal Anesthesia; Hemodynamics
MeSH Terms: interventions — Ondansetron; Injections

STUDY DESIGN:
Intervention Model Description: Ondansetron group (group O): 8mg(10 ml) of Ondansetron administrated 5 minutes before spinal anesthesia control group (group C): saline solution 0,9%(10ml)
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: an anesthesia nurse ; not included in the analysis, verified the allocation and prepared the syringe fulled with ondansetron or saline solution
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ondansetron group (Active Comparator): Ondansetron 8Mg/4mL Injection: administration of a bolus of 8 mg intravenous Ondansetron diluted in 10 ml of saline solution (0,09%) 5 minutes before spinal anesthesia
  Interventions: Drug: Ondansetron 8Mg/4mL Injection
- control group (Placebo Comparator): administration of 10 ml of saline solution (0,09%) 5 minutes before spinal anesthesia
  Interventions: Drug: Ondansetron 8Mg/4mL Injection

INTERVENTIONS:
Drug: Ondansetron 8Mg/4mL Injection — investigators administrated intravenously Ondansetron 8 mg 5 minutes before spinal anesthesia.
  Other Names: OD-C/S

SUMMARY:
BACKGROUND:

Spinal anesthesia (SA) induced maternal hypotension is the most frequent and troublesome complication in cesarean section (CS), compromising both maternal and neonatal well-being. Many strategies have been used to prevent its occurrence but no single technique has been confirmed to be completely effective. the investigators hypothesized that ondansetron, a serotonin-receptor-antagonist, could have beneficial effects on maternal hemodynamics during CS under SA.

METHODS:

In this prospective double-blind placebo-controlled study, one hundred healthy parturients were randomized to receive either 8 mg of intravenous ondansetron (group O) or the same volume of saline (group S), 5 minutes prior to the induction of SA. All women received a coloading volume of 500 ml of saline. Maternal hemodynamics: blood pressure, heart rate and cardiac output (CO) were measured with a non-invasive device based on pulse wave transit time: the esCCO device Nihon Kohden hemodynamic monitor. Ephedrine was administered to treat hypotension (systolic blood pressure less than 80% of baseline).

DETAILED DESCRIPTION:
1. Type of the study:

   After institutional ethical committee approval, we conducted a prospective double-blind, placebo-controlled, randomized study, at the department of anesthesiology of the Mahdia's university hospital, from August to November 2017.
2. Inclusion criteria:

   Parturients eligible for the present study are women who:

   are scheduled for elective cesarean section under spinal anesthesia. aged between 20 to 40 years. are with an American Society of Anesthesiologist (ASA) physical status of I-II are with a normal liver and renal function and fetal screening, and with no medical history of heart disease.

   are with a single fetus.
3. Protocol description:

3.1. Pre-operative time: A pre-anesthetic consultation, carried out at least 48 hours before the surgical procedure, made it possible to define eligible women for our study, to inform the parturients about the nature and the progress of the protocol and to collect their consent. Women were fasted for 6 hours before surgery and did not receive any premedication. In the morning of the intervention, a preoperative visit allowed us to check the application of instructions and the absence of intercurrent event.

3.2. per-operative time:

Randomization was performed at the entrance to the operating room after verification of the inclusion and exclusion criteria. All participants were randomly assigned to one of two groups according to a randomization table.

In the operating room, baseline values of noninvasive blood pressure (BP), electrocardiogram (ECG), and pulse oximetry (SPO2) were recorded using a Nihon Kohden monitor which also allowed a continuous non-invasive estimation of cardiac output (esCCO), based on pulse wave transit time (PWTT) which is automatically computed from pulse Oximetry waveform and electrocardiogram signals. After inputting the date of birth, sex, weight and height, the monitor was calibrated by the heart rate, pulse pressure, and PWTT.

Peripheral venous access was secured with an 18-gauge canula. An anesthesia nurse ; not included in the analysis ;verified the allocation and prepared the appropriate dose of Ondansetron (8 mg) with 0.9% saline solution to a total volume of 10 ml or a placebo of 0.9% saline solution10 ml. The syringes had no identifying markers indicating group allocation. The nurse injected the contents of the syringe intravenously over 60 s, 5 min before the lumbar puncture was performed. The anesthetist caring for the woman was blinded to group allocation.

Spinal anesthesia was induced in the sitting position at the L3-4 or L4-5 interspace, with a 25-gauge spinal needle pencil point. We administered 10 mg of 0.5% hyperbaric Bupivacaine, with 5ɤof Sufentanil and 100ɤof morphine. After injection, patients were immediately placed supine with 15 degrees left tilt. All women were rapidly coloaded with 500 ml of 0.9% saline solution.

Hemodynamic data were recorded at 2-min interval in the first 15-min and then every 5-min until the end of the procedure.

Sensory block height level was checked by assessing the perception of coldness using an alcohol swab, and motor block using Bromage scale.

Supplemental oxygen was administered via nasal canula at 2L/min. Maintenance fluids (10 ml/kg in the first one hour and 5ml/kg in the subsequent hours) were given at room temperature. Oxytocin was given following delivery of the fetus (5 IU directly and 10 IU in 250 ml of Glucose solution 5%). Antibioprophylaxis using 2g of Cefazolin was administered intravenously, in case of allergy, we used Clindamycin.

Neonatal Apgar score was noted at 1 and 5min after delivery.

Hypotension was defined as a decrease in systolic blood pressure (SBP)> 25% of baseline, and severe hypotension was defined as SBP< 80 mmHg. Treatment was initiated with intravenous Ephedrine 9 mg. More bolus of Ephedrine can be required.

Bradycardia, defined as a decrease in heart rate (HR) to less than 50 beats/min, was treated with intravenous atropine 0.5 mg.

Tachycardia was defined as HR >120 beats/min. Low flow was defined as a decrease in cardiac output (CO) > 15% from baseline.

3.3. Post-operative time:

After surgery, all parturients were transferred to the post-intervention monitoring room.

Standard monitoring of all parturients systematically included heart rate (HR), non invasive blood pressure (NIBP), respiratory frequency (RR), uterine globe tonus, bleeding, diuresis and temperature.

A glucose solution 5 % infusion enriched with electrolytes and comprising 20 IU of Oxytocin was instituted at a rate of 2 liters to 3l/24 h depending on the weight of the parturient.

The protocol of postoperative analgesia is ensured by the administration of Paracetamol in slow intravenous infusion at the dose of 1gevery 6 hours and Nefopam at the dose of 20 mg in slow infusion of 30 min every 8 hours. The postoperative prescription included also for all parturients Enoxaparin-based thrombophylaxis for 7 days.

ELIGIBILITY:
Inclusion Criteria:

Parturients eligible for the present study are women who:

* are scheduled for elective cesarean section under spinal anesthesia
* aged between 20 to 40 years
* are with an American Society of Anesthesiologist (ASA) physical status of I-II
* are with a normal liver and renal function and fetal screening, and with no medical history of heart disease.
* are with a single fetus.

Exclusion Criteria:

* Refusal to participate.
* Contraindication to spinal anesthesia
* Age <20 or >40 years.
* Obesity (body mass index (BMI) at term >35 kg/m2).
* History of hypersensitivity to study's drugs.
* History of long QT syndrome
* Hypertensive disorders of pregnancy.
* Women receiving selective serotonin reuptake inhibitors or migraine medications.
* Urgent cesarean section.
* Multiple pregnancies.
* Failure of spinal anesthesia.
* Conversion to general anesthesia.
* The occurrence of an anesthetic or surgical complication.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
hypotension | 5 min after spinal anesthésia
  decrease of systolic blood pressue with more than 25% from baseline values

SECONDARY OUTCOMES:
escco | 5 min after spinal anesthésia
  decrease of cardiac output (contious non invasive estimation of cardiac output based on pulse wave transit time) with more than 15% from baseline values
ephedrine consumption | during 2 hours of anesthetic time
  ephedrine dose used in perioperative time

CONTACTS AND LOCATIONS:
Overall Officials: bechir haddad, professor, Study Director — tunisian Ministry of Health
Locations (2):
- Tunisia (2):
  - Mahdia University Hospital, Mahdia
  - Ministry of Health, Tunis

IPD SHARING:
Plan to Share IPD: No